CLINICAL TRIAL: NCT02912169
Title: An Open-label, Non-Randomized, Multi-Center Study to Assess the Safety and Effects of Autologous Adipose-Derived Stromal Vascular Fraction (AD-SVF) Cells Delivered Intravenous (IV) and Intranasal in Patients With Alzheimer's Disease
Brief Title: Study to Assess the Safety and Effects of Autologous Adipose-Derived Stromal Cells in Patients With Alzheimer's Disease
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: company dissolved
Sponsor: Ageless Regenerative Institute (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AD-US-ALZ-001
Record Dates: First submitted 2016-04-06; First posted 2016-09-23 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Alzheimer's; Stem cell; Adipose-derived stem cells; ASC; ADSC
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous Adipose-derived Stromal Vascular Fraction infusion (Experimental): Autologous Adipose-derived Stromal Vascular Fraction (AD-SVF infusion) intravenous (IV) and Intranasal.
  Interventions: Procedure: Liposuction under local anesthesia; Biological: Infusion of AD-SVF via IV and Intranasal

INTERVENTIONS:
Procedure: Liposuction under local anesthesia — Procedure will be performed via liposuction to harvest Adipose-derived stromal vascular fraction cells.
  Other Names: Lipoaspiration; Adipose tissue harvesting
Biological: Infusion of AD-SVF via IV and Intranasal — IV and Intranasal Infusion of isolated AD-SVF

SUMMARY:
The intent of this clinical study is to answer the questions: 1) Is the proposed treatment safe and 2) Is treatment effective in improving the disease pathology of patients with Alzheimer's Disease and clinical outcomes?

DETAILED DESCRIPTION:
Autologous Adipose-derived Stromal Vascular Fraction (AD-SVF) will be infused intra-venous and Intra nasal. The therapy is composed of cells derived from a patients' own adipose tissue that are isolated within approximately 1 hour and immediately delivered back to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, age 55 or older
* Diagnosis of probable Alzheimer's disease, consistent with criteria from both: 1) National Institute of Neurological and Communicable Disease and Stroke and Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) and 2) Diagnostic and Statistical Manual of Mental Disorders (DSM IV)
* Up to date on all age and gender appropriate cancer screening per American Cancer Society (Refer to section 9.3 for more details).

Exclusion Criteria:

* Females who are pregnant or nursing or females of childbearing potential who are unwilling to maintain contraceptive therapy for the duration of the study
* Life expectancy < 6 months due to concomitant illnesses.
* Exposure to any investigational drug or procedure within 1 month prior to study entry or enrolled in a concurrent study that may confound results of this study.
* Active infectious disease. For patients who have tested positive for HIV, HTLV, HBV, HCV, CMV (IgM > IgG) and/or syphilis ,then an expert will be consulted as to patient eligibility based on the patient's infectious status
* Any illness which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results
* Patients on chronic immunosuppressive transplant therapy
* Systolic blood pressure (supine) ≤90 mmHg;
* Resting heart rate > 100 bpm;
* Active clinical infection.
* Cerebrovascular accident within 6 months prior to study entry
* Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or who in the opinion of the investigator are not suitable to participate.
* History of cancer (other than non-melanoma skin cancer or in-situ cervical cancer) in the last five years.
* Patient or legal guardian if applicable us unwilling and/or not able to give written informed consent.
* Dementia due to any condition other than AD, including vascular dementia

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Clinical Improvement in Mini Mental State Examination (MMSE) | Six months after therapy
  Improvement in MMSE six months after therapy

SECONDARY OUTCOMES:
Adverse Event | One year after stem cell therapy
  The safety of adipose-derived stem cell injection will be evaluated by assessment of the frequency and nature of adverse events occurring during the study injection and up to the 12-months period following treatment.
Clinical Improvement in Functional Activities Questionnaire (FAQ) | Three and six months after therapy
Clinical Improvement in Activities of Daily Living Questionnaire (ADL) | Three and six months after therapy
Clinical Improvement in Geriatric Depression Scale (GDS) | Three and six months after therapy
Clinical Improvement in Mini Mental State Examination (MMSE) | Three months after therapy

CONTACTS AND LOCATIONS:
Overall Officials: Sharon McQuillan, MD, Principal Investigator — Ageless Regenerative Institute
Locations (1):
- Ageless Regenerative Institute LLC, Aventura, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided